CLINICAL TRIAL: NCT00149539
Title: Abuse Potential of Buprenorphine/Naloxone as a Function of Maintenance Dose of Buprenorphine/Naloxone
Brief Title: Abuse Potential of Buprenorphine/Naloxone
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding ended for the study
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Johns Hopkins University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-7; R01-08045-7; DPMC
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2007-07

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Buprenorphine/naloxone

SUMMARY:
Buprenorphine is a treatment for opioid dependence. Naloxone is given in addition to buprenorphine in order to limit the abuse potential that is commonly associated with buprenorphine. The purpose of this study is to determine the abuse potential of high doses of buprenorphine/naloxone in opioid dependent individuals.

DETAILED DESCRIPTION:
Buprenorphine, a mixed agonist-antagonist opioid (or partial agonist), is a safe and effective treatment for opioid dependence. However, there is concern that buprenorphine may be abused due to its high abuse potential. A sublingual buprenorphine/naloxone combination tablet may reduce the risk of abuse associated with buprenorphine alone. The purpose of this study is to determine the abuse potential of acute doses of buprenorphine/naloxone in individuals who are maintained on different daily doses of sublingual buprenorphine/naloxone.

Participants will be maintained on both low and high doses of buprenorphine/naloxone. They will be challenged with low- and high-dose injected buprenorphine/naloxone, as well as active and placebo controls at each maintenance dose. During study visits, physiologic, subjective, and psychomotor responses to challenge sessions will be monitored and compared to known pharmacologic effects of opioid drugs.

ELIGIBILITY:
Inclusion Criteria:

* Actively abusing illegal opioids
* Qualifies for opioid substitution treatment (e.g., methadone or buprenorphine), but not in active treatment at the time of study entry
* Meets DSM-IV criteria for opioid dependence

Exclusion Criteria:

* Significant medical problems (e.g., insulin dependent diabetes mellitus)
* Non-substance use psychiatric disorders (e.g., schizophrenia)
* Seeking substance abuse treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2004-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Opiate withdrawal | up to one day
opiate agonist symptoms | up to one day
physiologic measures | up to one day

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States